CLINICAL TRIAL: NCT04894630
Title: Epidemiology, Clinical Profile and Treatment Outcomes of Bacterial and Fungal Keratitis in Minia Governate, Egypt
Brief Title: Infective Keratitis in Minia Governate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Nabila Abdelhaleem Aboeleyoon Mabrouk, prinicipal investigator, Minia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 61519
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Infective Keratitis
Keywords: infective keratitis; Bacterial keratitis; Fungal keratitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- infective keratitis (Other): 150 patients with mean age 30 (range 12 to 85 years), 90 patients (60 %) were males and 60 (40%) were females, clinically diagnosed as infective corneal ulcer, attending the Ophthalmology Department - Faculty of Medicine. Minia University, Minia, Egypt. From 2018 to 2020.
  Interventions: Other: antimicrobial treatment

INTERVENTIONS:
Other: antimicrobial treatment — Detailed history taking and all clinical findings were collected. Corneal scrapings were obtained from patients and subjected to staining and culture for bacterial and fungal pathogens; Bacterial and fungal growth were identified by standard laboratory procedures.

SUMMARY:
The purpose of the study is to determine the microbiological aetiology, epidemiological factors, and clinical profile and treatment outcomes of infective keratitis in Ophthalmology department, Minia University. Egypt

DETAILED DESCRIPTION:
Prospective, non-randomized, observational clinical series of cases, including 150 patients clinically diagnosed as infective corneal ulcer, attending the Ophthalmology Department - Faculty of Medicine. Minia University, Minia, Egypt. From 2018 to 2020.

Detailed history taking and all clinical findings were collected. Corneal scrapings were obtained from patients and subjected to staining and culture for bacterial and fungal pathogens; Bacterial and fungal growth were identified by standard laboratory procedures.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed as infective corneal ulcer, attending the Ophthalmology Department - Faculty of Medicine - Minia University, Minia, Egypt

Exclusion Criteria:

* healed keratitis

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Positive smear and culture | 1 month
  positive smear culture for bacteria and fungi

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelghany, ASS PROF, Study Director — Minia University
Locations (1):
- Minia University, Minya, Egypt

REFERENCES:
- [Derived] Mabrouk NA, Abdelkader MF, Abdelhakeem MA, Mourad KM, Abdelghany AA. Epidemiology, clinical profile and treatment outcomes of bacterial and fungal keratitis. Int Ophthalmol. 2022 May;42(5):1401-1407. doi: 10.1007/s10792-021-02128-x. Epub 2021 Nov 28. PMID 34839447